CLINICAL TRIAL: NCT07039955
Title: Effectiveness of Daily Chlorhexidine Bathing and Antibiotic and Proton Pump Inhibitor (PPI) Stewardship in Preventing Transmission and Infection Caused by Carbapenemase-Producing Enterobacteriaceae (CPE)
Brief Title: Effect of Daily Chlorhexidine Bathing and Antibiotic/PPI Stewardship on Prevention of CPE Transmission and Infection
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Wonju Severance Christian Hospital (Other); Gangneung Asan Hospital (Other); National Institute of Health, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2025-05-001
Record Dates: First submitted 2025-06-06; First posted 2025-06-26 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Carbapenemase-Producing Enterobacteriaceae (CPE); Healthcare-Associated Infections (HAIs)
Keywords: Carbapenemase-Producing Enterobacteriaceae; Healthcare-Associated Infections; Intensive Care Unit; infection control; Daily Chlorhexidine Bathing; Antimicrobial Stewardship; Proton Pump Inhibitor Stewardship; Chlorhexidine (CHG) Skin Concentration; Chlorhexidine (CHG) Minimum Inhibitory Concentration (MIC)
MeSH Terms: conditions — Cross Infection | interventions — Anti-Infective Agents

STUDY DESIGN:
Intervention Model Description: Cluster-randomized crossover trial involving six intensive care units (ICUs) across three university-affiliated hospitals. Each hospital contributes two ICUs, which are randomized to either the intervention or control group for six months, followed by crossover to the opposite group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHG Bathing + Antimicrobial/PPI Stewardship (Experimental): Patients admitted to intensive care units (ICUs) assigned to the intervention group will receive daily bathing using no-rinse, 4% chlorhexidine gluconate (CHG)-impregnated washcloths. In addition, targeted antimicrobial stewardship focused on reducing unnecessary carbapenem use and PPI stewardship aimed at limiting inappropriate PPI prescriptions will be implemented.
  Interventions: Behavioral: Daily Chlorhexidine Bathing; Behavioral: Antimicrobial and PPI Stewardship Program
- Standard Bathing + Antimicrobial/PPI Stewardship (Active Comparator): Patients admitted to ICUs assigned to the control group will receive standard daily bathing without chlorhexidine. The same antimicrobial and PPI stewardship interventions applied in the intervention group will also be implemented in the control group.
  Interventions: Behavioral: Antimicrobial and PPI Stewardship Program; Behavioral: Standard Bathing

INTERVENTIONS:
Behavioral: Daily Chlorhexidine Bathing — Daily bathing using no-rinse, 4% chlorhexidine gluconate (CHG)-impregnated washcloths will be implemented in ICUs assigned to the intervention group. The purpose is to reduce CPE colonization and infection by maintaining effective residual CHG skin concentrations. Bathing will be performed by trained nursing staff following standardized protocols.
  Arms: CHG Bathing + Antimicrobial/PPI Stewardship
Behavioral: Antimicrobial and PPI Stewardship Program — A targeted stewardship program will be implemented to reduce unnecessary carbapenem use and inappropriate proton pump inhibitor (PPI) prescriptions. The program includes audit and feedback, education of ICU physicians, and monthly monitoring of antimicrobial and PPI usage. Stewardship activities will be uniformly applied across both intervention and control ICUs.
Behavioral: Standard Bathing — Patients in ICUs assigned to the control group will receive standard daily bathing without the use of chlorhexidine. No CHG-containing products will be applied. This represents usual care in the participating hospitals.
  Arms: Standard Bathing + Antimicrobial/PPI Stewardship

SUMMARY:
This multicenter, cluster-randomized crossover trial aims to evaluate the effectiveness and safety of a bundled intervention-including daily chlorhexidine bathing and targeted antimicrobial and proton pump inhibitor (PPI) stewardship-for preventing colonization and infection caused by carbapenemase-producing Enterobacteriaceae (CPE) in intensive care units (ICUs) across three university-affiliated hospitals in South Korea.

Each hospital will include two ICUs, randomized to either the intervention or control group for six months, followed by a crossover. The intervention group will receive daily bathing using no-rinse, 4% chlorhexidine gluconate (CHG)-impregnated washcloths along with antimicrobial and PPI stewardship focused on reducing unnecessary carbapenem and PPI use. The control group will receive standard bathing without chlorhexidine, while receiving the same stewardship interventions as the intervention group.

Primary outcomes include the incidence and prevalence of CPE colonization and CPE-attributable healthcare-associated infections such as bloodstream infections, hospital-acquired pneumonia, and urinary tract infections. Secondary outcomes include evaluation of residual CHG skin concentrations, comparison with CHG minimum inhibitory concentrations (MICs) of CPE isolates, impact of feedback on adherence to bathing protocols, and assessment of adverse skin reactions to CHG bathing.

Findings from this study are expected to provide evidence-based guidance on the effectiveness and feasibility of combining daily chlorhexidine bathing with no-rinse, 4% CHG-impregnated washcloths and stewardship interventions to control the spread of CPE in high-risk healthcare settings.

DETAILED DESCRIPTION:
Carbapenemase-producing Enterobacteriaceae (CPE) are a critical public health threat, particularly in healthcare settings where vulnerable patients are at increased risk of colonization and infection. In South Korea, the number of reported CPE cases has increased sharply in recent years, necessitating the implementation of high-impact, evidence-based strategies for prevention and control.

This multicenter, cluster-randomized crossover trial is being conducted in six intensive care units (ICUs) across three university-affiliated hospitals in South Korea. The primary aim of the study is to evaluate the effectiveness and safety of a bundled intervention consisting of daily chlorhexidine bathing and targeted antimicrobial and proton pump inhibitor (PPI) stewardship in reducing CPE colonization and infection.

Each participating hospital will contribute two ICUs. One ICU will initially serve as the intervention unit and the other as the control unit for six months, after which the roles will be crossed over for an additional six months. The intervention group will receive daily bathing using no-rinse, 4% chlorhexidine gluconate (CHG)-impregnated washcloths, along with antimicrobial and PPI stewardship interventions focused on reducing unnecessary use of carbapenems and PPIs. The control group will receive standard bathing without chlorhexidine, while receiving the same stewardship measures as the intervention group.

Primary outcomes include the incidence and prevalence of CPE colonization and CPE-attributable healthcare-associated infections (HAIs), such as bloodstream infections, hospital-acquired pneumonia, and urinary tract infections. Surveillance cultures will be obtained per institutional protocols and national guidelines, including rectal swabs at ICU admission and weekly thereafter.

Secondary outcomes include:

1. Assessment of residual CHG skin concentrations at 3-month intervals using standardized skin swabs and comparison of these concentrations with the minimum inhibitory concentrations (MICs) of CPE isolates obtained from clinical and surveillance cultures to evaluate the adequacy of chlorhexidine exposure.
2. Evaluation of adherence to CHG bathing protocols through quarterly feedback of CHG skin concentration results to ICU staff.
3. Assessment of adverse skin reactions associated with CHG bathing to evaluate its safety in critically ill patients.

Skin swab samples will be obtained from the neck, axilla, and groin using a standardized technique. CHG concentrations will be analyzed via a semiquantitative colorimetric assay. CPE isolates will undergo broth microdilution testing to determine the MICs of CHG, following modified Clinical and Laboratory Standards Institute (CLSI) guidelines. CPE isolates will undergo broth microdilution MIC testing based on modified CLSI guidelines.

In parallel, antimicrobial and PPI utilization will be monitored using antibiotic use density (AUD) metrics. Stewardship interventions will focus on minimizing unnecessary use of carbapenems and PPIs, particularly for ventilator-associated pneumonia prophylaxis, and promoting use of alternatives where appropriate. Monthly trends in AUDs will be tracked for carbapenems, ampicillin/sulbactam, ceftazidime/avibactam, cefiderocol, colistin, and other key antibiotics, as well as PPIs and H2 blockers.

This study is designed to provide high-quality evidence on the effectiveness and feasibility of bundled interventions for the prevention of CPE transmission and infection in high-risk ICU settings. Findings from this trial may inform national infection control guidelines and support the broader implementation of CHG-based decolonization and stewardship strategies in similar healthcare environments.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older
2. Admitted to one of the participating intensive care units (ICUs):

   * Chuncheon Sacred Heart Hospital: CICU or NCU
   * Wonju Severance Christian Hospital: MICU or NSICU
   * Gangneung Asan Hospital: MICU or SICU

Exclusion Criteria:

1. Age 18 years or younger
2. Patients with extensive burns
3. Patients with a known hypersensitivity to chlorhexidine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5760 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of CPE Colonization and Infection | From ICU admission up to ICU discharge (an average of 10-14 days)
  Incidence of new colonization or infection with carbapenemase-producing Enterobacteriaceae (CPE) during ICU admission, confirmed through active surveillance cultures (e.g., rectal swab) and clinical diagnostic specimens (e.g., blood, respiratory, or urine cultures).
  Infections will be defined according to CDC/NHSN criteria for healthcare-associated infections.

SECONDARY OUTCOMES:
Residual CHG Skin Concentration vs. CPE MIC Comparison | Measured at 3-month intervals during intervention periods
  Assessment of residual skin concentrations of chlorhexidine gluconate (CHG) using standardized skin swabs, and comparison with the minimum inhibitory concentrations (MICs) of CPE isolates obtained from clinical or surveillance cultures to determine adequacy of CHG exposure.
Proportion of CHG Bathing Days Adherent to Protocol Based on CHG Skin Concentration, Checklist Compliance, and EMR Audit | Approximately Day 15 of Months 0, 3, and 6 during the intervention period
  This outcome assesses adherence to the daily chlorhexidine gluconate (CHG) bathing protocol among ICU patients. Adherence will be evaluated using a combination of:
  1. Colorimetric CHG skin concentration testing, with adherence defined as CHG concentration ≥125 µg/mL on at least 2 of 3 body sites;
  2. Chlorhexidine Bathing Checklist completed by bedside staff; and
  3. Electronic Medical Record (EMR) audit for daily documentation of CHG bathing.
  Feedback on adherence results will be provided to ICU staff, and its impact on improving adherence rates will be evaluated.
Incidence of Adverse Skin Reactions Related to CHG Bathing | Daily during the intervention period, from ICU admission up to ICU discharge (an average of 10-14 days)
  Monitoring and reporting of adverse skin reactions (e.g., erythema, rash, itching, blistering) associated with daily chlorhexidine bathing using 4% CHG-impregnated washcloths. Skin assessments will be conducted by trained staff through direct observation and chart review.
Monthly Trends in Antimicrobial and PPI Use | Monthly, from intervention start (Month 1) to study end (Month 12)
  Monthly analysis of antimicrobial and PPI utilization, measured as days of therapy (DOT) per 1,000 patient-days, including carbapenems, ampicillin/sulbactam, ceftazidime/avibactam, cefiderocol, and PPI vs. H2 blocker use.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Chuncheon Sacred Heart Hospital, Hallym University College of Medicine, Chuncheon, Gangwon-do
  - Gangneung Asan Hospital, University of Ulsan College of Medicine, Gangneung, Gangwon-do
  - Wonju Severance Christian Hospital, Yonsei University Health System, Wŏnju, Gangwon-do

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy concerns and the nature of the cluster-level intervention design.

REFERENCES:
- [Background] Rhee Y, Hayden MK, Schoeny M, Baker AW, Baker MA, Gohil S, Rhee C, Talati NJ, Warren DK, Welbel S, Lolans K, Bahadori B, Bell PB, Bravo H, Dangana T, Fukuda C, Habrock Bach T, Nelson A, Simms AT, Tolomeo P, Wolf R, Yelin R, Lin MY; CDC Prevention Epicenters Program. Impact of measurement and feedback on chlorhexidine gluconate bathing among intensive care unit patients: A multicenter study. Infect Control Hosp Epidemiol. 2023 Sep;44(9):1375-1380. doi: 10.1017/ice.2023.177. Epub 2023 Sep 13. PMID 37700540
- [Background] Willems RPJ, van Dijk K, Ket JCF, Vandenbroucke-Grauls CMJE. Evaluation of the Association Between Gastric Acid Suppression and Risk of Intestinal Colonization With Multidrug-Resistant Microorganisms: A Systematic Review and Meta-analysis. JAMA Intern Med. 2020 Apr 1;180(4):561-571. doi: 10.1001/jamainternmed.2020.0009. PMID 32091544
- [Background] Rhee Y, Simms AT, Schoeny M, Baker AW, Baker MA, Gohil S, Rhee C, Talati NJ, Warren DK, Welbel S, Lolans K, Bell PB, Fukuda C, Hayden MK, Lin MY; CDC Prevention Epicenters Program. Relationship between chlorhexidine gluconate concentration and microbial colonization of patients' skin. Infect Control Hosp Epidemiol. 2024 May 28:1-6. doi: 10.1017/ice.2024.81. Online ahead of print. PMID 38804007
- [Background] Patel A, Parikh P, Dunn AN, Otter JA, Thota P, Fraser TG, Donskey CJ, Deshpande A. Effectiveness of daily chlorhexidine bathing for reducing gram-negative infections: A meta-analysis. Infect Control Hosp Epidemiol. 2019 Apr;40(4):392-399. doi: 10.1017/ice.2019.20. Epub 2019 Feb 26. PMID 30803462
- [Background] Climo MW, Yokoe DS, Warren DK, Perl TM, Bolon M, Herwaldt LA, Weinstein RA, Sepkowitz KA, Jernigan JA, Sanogo K, Wong ES. Effect of daily chlorhexidine bathing on hospital-acquired infection. N Engl J Med. 2013 Feb 7;368(6):533-42. doi: 10.1056/NEJMoa1113849. PMID 23388005